CLINICAL TRIAL: NCT00623545
Title: Bioenergetic Alterations After Exenatide Administration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2007-0235
Record Dates: First submitted 2008-02-14; First posted 2008-02-26 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: Exenatide; Byetta; weight loss; energy expenditure; normal volunteers
MeSH Terms: conditions — Weight Loss | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exenatide (Experimental): Exenatide. Dose was 5 microgram for 2 weeks that was increased to 10 microgram for 10 weeks Each subject serves as their own control for outcome measures taken before and during drug treatment.
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — Exenatide dose was 5 microgram for 2 weeks that was increased to 10 microgram for 10 weeks of treatment.
  Other Names: Byetta

SUMMARY:
The purpose of this study is to find out how exenatide causes weight loss. Specifically, the study is assessing how exenatide may change how people take in energy (energy intake), as well as how it may effect how people use energy (energy expenditure).

DETAILED DESCRIPTION:
The bioenergetics study is looking at how and why the diabetes drug exenatide causes people to lose weight.Bioenergetics is the study of how your body burns calories.

Adults 18-65 who do not have diabetes and have a body mass index (BMI) between 30 and 40 may be eligible. Women who could get pregnant must be on birth control during the study and women who are pregnant cannot participate in the study.

Subjects will take exenatide for 12 weeks. There are 6 study visits in the Univ. Wisconsin Hospital General Clinical Research Center. Visits range from 1 to 6 hours and include blood and urine tests, resting metabolic rate testing over a four hour period, physical exam, ECG, and a be bone mineral density testing at another clinic during 2 clinic visits of the study.

All study procedures and testing are free of charge.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* BMI between 30 and 40 kg/m2
* Women with a negative pregnancy test at baseline, who are sterile, using contraceptives or in a committed relationship with someone who is sterile or using contraception
* Absence of weight change greater than 3 kg in the previous 6 months

Exclusion Criteria:

* Women who are pregnant or lactating
* Current or recent (6 months) enrollment in a commercial or self prescribed weight loss or exercise program
* Use of weight loss medication
* A history of metabolic disease i.e. renal, endocrine, hepatic or gastrointestinal disease that would impact the outcome of the study
* Presence of medical conditions that are known to affect energy expenditure (i.e. hyperthyroidism, rheumatoid arthritis, AIDS among others)
* History of hypoglycemia
* A history of psychiatric or eating disorder
* Abnormal EKG
* Previous history of pancreatitis
* Previous history of gastroparesis or GI motility disorder
* Use of medications that can affect GI motility
* History of organ transplantation
* Other comorbid conditions which may preclude the subject's ability to complete the study
* Use of a carbonic anhydrase inhibitor such as acetazolamide

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Bradley, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Univ Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Result] Bradley DP, Kulstad R, Schoeller DA. Exenatide and weight loss. Nutrition. 2010 Mar;26(3):243-9. doi: 10.1016/j.nut.2009.07.008. PMID 20152707
- [Derived] Bradley DP, Kulstad R, Racine N, Shenker Y, Meredith M, Schoeller DA. Alterations in energy balance following exenatide administration. Appl Physiol Nutr Metab. 2012 Oct;37(5):893-9. doi: 10.1139/h2012-068. Epub 2012 Jun 26. PMID 22735035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was ca. 5/1/2008 to 6/30/2010. Subjects were recruited through local advertisements
Pre-assignment Details: Subjects were not entered if they failed to meet entry criteria or failed to attend informational appointment
Groups:
- Single Arm Study of Exenatide Treatment: Subjects serve as their own controls. Measures of outcome variables are made before treatment and again at the end of the1 treatment period made. Outcomes are based on the change in these variables.
Period: Overall Study
Arm/Group | Single Arm Study of Exenatide Treatment
Started | 28
Completed | 18
Not Completed | 10
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Groups:
- Single Arm Study of Exenatide Treatment: Subjects serve as their own controls. Measures of outcomes are performed before and at the end of treatment. Outcomes are based on the change in the variables.
Arm/Group | Single Arm Study of Exenatide Treatment
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in Energy Intake Measured Before Treatment and at the End of Treatment.
Description: Energy intake is as calculated from energy expenditure as measured by doubly labeled water and change in body energy stores before and at the end of treatment. Units are kcal/d.
Time Frame: 3 months
Population: Those that completed baseline and final measurements.
Measure: Mean (Standard Deviation); unit: kcal/d
Groups:
- Exenitide Treatment: There is one treatment arm. Subjects serve as their own controls for the outcome measure. The measures are made before the treatment is started at during the end of the treatment.
Arm/Group | Exenitide Treatment
Number analyzed (Participants) | 18
kcal/d | -167 (173)
Statistical Analysis 1: Comparison: Exenitide Treatment; Previously published literature showed an average weight loss of 1.8 kg at 12 weeks of exenatide treatment. This was converted to differ- ence in TEE, estimating an average imbalance of 2 kg × 7800 kcal·kg-1 divided by 84 days or 185 kcal·day-1.We demonstrated an average reproducibility of the DLW method of 6% or 240 kcal·day-1. For a 5% probability of finding this difference with a power of 80%, we determined a need for 14 subjects to complete the study; Test type: Superiority or Other; p = 0.001, ANOVA — The a prior threshold for statistical significance was p< 0.05; Mean Difference (Net) = 185, Standard Deviation 240 — units are kcal/d
Statistical Analysis 2: Comparison: Exenitide Treatment; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0

2. Secondary Outcome: Weight Loss After Administration of Exenatide.
Description: Body weight after overnight fast in light clothing
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Exenitide Treatment
Number analyzed (Participants) | 18
kg | -2.0 (2.8)
Statistical Analysis 1: Comparison: Exenitide Treatment; The null hypothesis was that energy intake was unchanged between the period before treatment and at the end of treatment; Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Exenitide Treatment; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: periodic self-report
Arm/Group | Single Arm Study of Exenatide Treatment
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 6/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Study of Exenatide Treatment (N=28)
nausea (Gastrointestinal disorders) | 5 (5)
claustrophobia (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
study was limited by the number of subjects who did not complete the study as a result of nausea. The nausea was short-lived and mild in all subjects that completed the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No